CLINICAL TRIAL: NCT05200923
Title: Pelvic Health Electrically Evoked Recording (PEER) 2 Study
Acronym: PEER 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MDT20063
Record Dates: First submitted 2021-12-20; First posted 2022-01-21 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Overactive Bladder; Fecal Incontinence; Urinary Retention
MeSH Terms: conditions — Urinary Bladder, Overactive; Fecal Incontinence; Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Pelvic health Electrically Evoked Recording (PEER) 2 Study (Experimental): Collect physiological signals
  Interventions: Device: Sacral Neuromodulation

INTERVENTIONS:
Device: Sacral Neuromodulation — Sacral neuromodulation delivers electrical stimulation to a sacral nerve

SUMMARY:
To collect physiological signals at several timepoints during the therapy evaluation period.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this non-applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.)

ELIGIBILITY:
Inclusion Criteria:

Overactive Bladder Criteria Inclusion Criteria

1. 18 years of age or older
2. Candidate for or undergoing Medtronic InterStim lead implant for labeled indication* requiring an advanced evaluation
3. Willing and able to provide signed and dated informed consent
4. Willing and able to independently and accurately complete diaries, questionnaires, attend visits, and comply with the study protocol
5. Willing to maintain current regimen (dosage and frequency) of any OAB medication from baseline diary through the end of therapy evaluation
6. For subjects with urinary urge incontinence, have a diagnosis of OAB as demonstrated on a voiding diary by having a minimum of 3 episodes of urinary urge incontinence in the first 72 hours (Episodes must have a mild, moderate, or severe degree of urgency to meet this criterion) of the voiding diary.
7. For subjects with urinary frequency, have a diagnosis of OAB as demonstrated on a voiding diary with greater than or equal to 8 urgency frequency episodes per day within the first 72 hours of the voiding diary.

Note*: Candidate for or undergoing a Medtronic InterStim lead implant for labeled indication means that a clinical decision has already been made between a physician and the patient to undergo Medtronic Interstim lead implant to treat the subject's condition. This decision is to be made prior to discussing with the patient whether to enroll in the study.

Non-Obstructive Urinary Retention Inclusion Criteria

1. 18 years of age or older
2. Candidate for or undergoing Medtronic InterStim lead implant for labeled indication* requiring an advanced evaluation
3. Willing and able to provide signed and dated informed consent
4. Willing and able to independently and accurately complete diaries, questionnaires, attend visits, and comply with the study protocol
5. Willing to maintain current regimen (dosage and frequency) of any NOUR medication from baseline diary through the end of therapy evaluation
6. Have a diagnosis of non-obstructive urinary retention with an elevated postvoid residual (PVR) that has persisted for at least six months and is documented on two or more separate occasions.

Note*: Candidate for or undergoing a Medtronic InterStim lead implant for labeled indication means that a clinical decision has already been made between a physician and the patient to undergo Medtronic Interstim lead implant to treat the subject's condition. This decision is to be made prior to discussing with the patient whether to enroll in the study.

Fecal Incontinence Inclusion Criteria

1. 18 years of age or older
2. Candidate for or undergoing Medtronic InterStim lead implant labeled indication* requiring an advanced evaluation
3. Willing and able to provide signed and dated informed consent
4. Willing and able to independently and accurately complete diaries, questionnaires, attend visits, and comply with the study protocol
5. Willing to maintain current regimen (dosage and frequency) of any FI medication from baseline diary through the end of therapy evaluation
6. Have a diagnosis of fecal incontinence as demonstrated by 3-day a bowel diary as greater than or equal to 1 incontinent episode of more than staining (i.e., either slight, moderate, or severe soiling)

Note*: Candidate for or undergoing a Medtronic InterStim lead implant for labeled indication means that a clinical decision has already been made between a physician and the patient to undergo Medtronic Interstim lead implant to treat the subject's condition. This decision is to be made prior to discussing with the patient whether to enroll in the study.

Exclusion Criteria:

Overactive Bladder Criteria Exclusion Criteria

1. Currently enrolled or planning to enroll in an interventional clinical study that could potentially confound the study results (co-enrollment in an interventional study is only allowed when documented pre-approval is obtained from the Medtronic study manager or designee)
2. Implanted with a neurostimulator, pacemaker or defibrillator
3. Pelvic floor muscle dysfunction due to surgical intervention or injury
4. Have neurological conditions such as multiple sclerosis, clinically significant peripheral neuropathy or spinal cord injury (e.g., paraplegia)
5. History of diabetes unless the diabetes is well-controlled through diet and/or medications
6. Have symptomatic urinary tract infection (UTI)
7. Have primary stress incontinence or mixed incontinence where the stress component overrides the urge component
8. Treatment of voiding behavior with botulinum toxin in the past 9 months or any plan to have botulinum toxin treatment during the study
9. Treatment of symptoms with tibial neuromodulation therapy in the last 3 months
10. Have knowledge of planned magnetic resonance imaging (MRIs) during the therapy evaluation portion of the study
11. Have knowledge of planned shortwave diathermy, microwave diathermy, or therapeutic diathermy
12. Women who are pregnant or planning to become pregnant
13. Current urinary tract mechanical obstruction (e.g. benign prostatic enlargement or urethral stricture)
14. Characteristics indicating a poor understanding of the study or characteristics that indicate the subject may have poor compliance with the study protocol requirements

Non-Obstructive Urinary Retention Exclusion Criteria

1. Currently enrolled or planning to enroll in an interventional clinical study that could potentially confound the study results (co-enrollment in an interventional study is only allowed when documented pre-approval is obtained from the Medtronic study manager or designee)
2. Implanted with a neurostimulator, pacemaker or defibrillator
3. Pelvic floor muscle dysfunction due to surgical intervention or injury
4. Have neurological conditions such as multiple sclerosis, clinically significant peripheral neuropathy or spinal cord injury (e.g., paraplegia)
5. History of diabetes unless the diabetes is well-controlled through diet and/or medications
6. Have symptomatic urinary tract infection (UTI)
7. Treatment of symptoms with tibial neuromodulation therapy in the last 3 months
8. Have knowledge of planned magnetic resonance imaging (MRIs) during the therapy evaluation portion of the study
9. Have knowledge of planned shortwave diathermy, microwave diathermy, or therapeutic diathermy
10. Women who are pregnant or planning to become pregnant
11. Current urinary tract mechanical obstruction (e.g. benign prostatic enlargement or urethral stricture)
12. Characteristics indicating a poor understanding of the study or characteristics that indicate the subject may have poor compliance with the study protocol requirements

Fecal Incontinence Exclusion Criteria

1. Currently enrolled or planning to enroll in an interventional clinical study that could potentially confound the study results (co-enrollment in an interventional study is only allowed when documented pre-approval is obtained from the Medtronic study manager or designee)
2. Implanted with a neurostimulator, pacemaker or defibrillator
3. Pelvic floor muscle dysfunction due to surgical intervention or injury
4. Have neurological conditions such as multiple sclerosis, clinically significant peripheral neuropathy or spinal cord injury (e.g., paraplegia)
5. Have uncorrected high grade internal rectal prolapse
6. Treatment of symptoms with tibial neuromodulation therapy in the last 3 months
7. Have knowledge of planned magnetic resonance imaging (MRIs) during the therapy evaluation portion of the study
8. Have knowledge of planned shortwave diathermy, microwave diathermy, or therapeutic diathermy
9. Women who are pregnant or planning to become pregnant
10. Characteristics indicating a poor understanding of the study or characteristics that indicate the subject may have poor compliance with the study protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2026-12-18 (Estimated); Study Completion 2026-12-18 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with physiological signals collected at each timepoint | 1 day to 7 months
  The proportion of subjects with evaluable signals will be summarized at each timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Peterson, Study Director — Medtronic Pelvic Health
Locations (7):
- United States (7):
  - Indiana University Health Methodist Research Institute, Indianapolis, Indiana
  - LSUHSC Department of Urology, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Mayo Clinic Urology/Urogynecology Department, Rochester, Minnesota
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - OhioHealth Physician's Group Urology, Hilliard, Ohio
  - DHR Health Institute for Research and Development, Edinburg, Texas

IPD SHARING:
Plan to Share IPD: No